CLINICAL TRIAL: NCT06097208
Title: BMI Development and Risk of Overweight and Obesity When Attending a Community-based Health Promotion and Obesity Prevention Intervention in Kindergartens
Brief Title: BMI Development and Risk of Overweight and Obesity in Children
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Healthy weight in kindergarten
Record Dates: First submitted 2023-10-03; First posted 2023-10-24 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Health Behavior; Child Obesity; Body Weight
Keywords: Obesity; Body Mass Index; Children; Kindergarten
MeSH Terms: conditions — Health Behavior; Pediatric Obesity; Body Weight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: Children who attended kindergartens actively delivering a community-based health promotion and obesity prevention intervention
  Interventions: Behavioral: community-based health promotion and obesity prevention intervention
- No-intervention Group: Children who attended usual care kindergartens

INTERVENTIONS:
Behavioral: community-based health promotion and obesity prevention intervention — The intervention involving measurements of children aged three- to four-years old in kindergartens, parents of the children had the opportunity of individual contact with a community health nurse, and education to kindergartens manager and employees e.g. pedagogues and kitchen staff. as well to parents of children in kindergartens.
  Groups: Intervention Group

SUMMARY:
The goal of this observational study is to investigate differences in attained BMI and the proportion of overweight/obesity at school entrance in children who attended kindergartens actively delivering a community-based health promotion and obesity prevention intervention compared to children who attended usual care kindergartens. Further questions it aims to answer are:

* Explore the prevalence of attainted overweight/obesity in children at six years of age, who attended kindergartens delivering intervention compared with usual care kindergartens.
* Explore the development of obesity, overweight and normal weight in children from three-, four- to six years of age, who attended kindergartens delivering intervention.

ELIGIBILITY:
Inclusion Criteria:

* All children with eligible information on one measure of BMI after school entrance

Exclusion Criteria:

* <7 years of age

Ages: 3 Years to 7 Years | Sex: All
Age Groups: Child
Study Population: The present study is based on data from a total of approximately 3000 children (six-year-olds) at school entrance in the period 2021-2022, of whom approximately 2000 children attended the community-based health promotion and obesity prevention intervention in kindergartens (intervention group), from Viborg Municipality, and approximately 1000 children attended usual care kindergarten (no-intervention group), from Skive Municipality, both municipalities located in The Central Denmark Region. Further, a subset of approximately 700 children from the intervention group have been measured with height and weight in kindergartens (three- to four-year-olds).
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
BMI after school entrance at 6 years of age | 2018-2023
  Differences in attained BMI after school entrance will be defined as weight and height combined to report BMI in kg/m^2 for sex and age.
Proportion of children with overweight/obesity at 6 years of age | 2018-2023
  The proportion of overweight/obesity after school entrance will be defined as weight and height combined to report BMI in kg/m^2 for sex and age. The proportion of overweight/obesity will be defined as BMIz≥1

IPD SHARING:
Plan to Share IPD: Undecided